CLINICAL TRIAL: NCT07022587
Title: A Bioresorbable Sirolimus-eluting scaﬀold Versus a Metallic Sirolimus-eluting Stent for the Treatment of de Novo Coronary Artery Lesions: a Randomized, Open-label, Non-inferiority Trial
Brief Title: Bioresorbable Sirolimus-eluting scaﬀold in de Novo Coronary Artery Lesions
Acronym: REC-CAGEFREE Ⅳ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the Department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20252116-C-1
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: De Novo Stenosis; Coronary Artery Disease
Keywords: bioresorbable vascular scaffold; drug-eluting stent; de novo stenosis; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioresorbable scaffold (BRS) (Experimental)
  Interventions: Device: Sirolimus-eluting bioresorbable scaffolds
- Drug-eluting stents (DES) (Active Comparator)
  Interventions: Device: Sirolimus-eluting stents

INTERVENTIONS:
Device: Sirolimus-eluting bioresorbable scaffolds — The Firesorb BRS (MicroPort Medical, Shanghai, China) is a balloon-expandable scaffold with a highly crystallized PLLA backbone, abluminally coated with a poly(D, L-lactide) (PDLLA) matrix incorporating sirolimus (4 μg/mm) through highly accurate and precise point spraying techniques. The scaffold thickness is 100 μm for devices with diameters of 2.5 and 2.75 mm, and 125 μm for those ranging from 3.0 to 4.0 mm in diameter. There are two radiopaque markers at each end of the scaffold, which can identify the position of the stent under X-ray monitoring and help to accurately locate the scaffold.
  Arms: Bioresorbable scaffold (BRS)
Device: Sirolimus-eluting stents — The Firehawk™ stent (MicroPort Medical, Shanghai, China) is a third-generation balloon-expandable L605 cobalt chromium stent with abluminal grooves containing a biodegradable polymer, which provides controlled release of the anti-proliferative medicinal substance sirolimus. The polymer is biodegradable, leaving only the metallic stent as a permanent implant. The stent is mounted on a rapid exchange delivery catheter system. The unique abluminal grooves are scored at the outer surface of the struts (total strut thickness: 86 μm), with an average sirolimus dosage of 3 µg/mm stent lengths.
  Arms: Drug-eluting stents (DES)

SUMMARY:
Bioresorbable scaffold (BRS) was designed aiming to avoid the late adverse events associated with permanent metallic stents by providing temporary support to the vessel wall and promoting vessel remodeling, plaque reduction, and restoring vasomotion after its full absorption. As the first FDA-approved BRS, ABSORB BRS was associated with a significantly higher risk of late scaffold thrombosis compared with everolimus-eluting stent (EES). As a result, the ESC-EAPCI task force recommended that the current ABSORB BRS should not be preferred over conventional DES in clinical practice. To solve this dilemma, improved scaffold technology and optimal implantation techniques are necessary.

The latest generation Firesorb BRS is a PLLA backbone scaffold system abluminally coated with poly(D, L-lactide) mixed with sirolimus using highly accurate and precise point spraying techniques. Compared to the ABSORB BRS, Firesorb features a thinner stent thickness (100-125 μm) while maintaining sufficient radial support, enabling faster degradation and a shorter duration of presence in the coronary. Additionally, inspired by the design of the Firehawk DES, its unique spot-coating process applies a single-sided coating layer exclusively to the stent's outer surface, enabling targeted drug release. Preclinical trials have demonstrated favorable performance for Firesorb, culminating in its approval by the National Medical Products Administration (NMPA) in 2024.

Against these backgrounds, we have designed this trial to investigate whether the Firesorb BRS is non-inferior to the drug-eluting stent in terms of the Device-Oriented Composite Endpoint (DoCE) in patients undergoing percutaneous coronary intervention for de novo lesions.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria

1. Patients with an indication for PCI due to acute or chronic coronary syndrome
2. Patients who understand the study's objectives, voluntarily participate, sign the informed consent form, and are willing to undergo regular follow-up

Angiographic inclusion criteria

1. De novo lesion(s)
2. Target vessel diameter of ≥ 2.5 mm to ≤ 4.00 mm, target lesion length ≤ 25 mm (visual estimation)
3. Target lesion is NOT

   1. Severely calcified
   2. In-stent restenosis
   3. Diffused lesion requiring stent overlapping or more than one stent
   4. Located in the left main, aorto-ostial, proximal LAD/LCX/RCA involving vessel ostia (stent coverage required within 3 mm of vessel ostia), surgical graft, myocardial bridge, or chronic total occlusion
   5. Bifurcation requiring two stents or involving a side branch that is ≥ 2.5 mm in diameter
   6. Located in the target vessel with severe tortuosity

Exclusion Criteria:

1. Age < 18 years, or > 75 years
2. Patient is a woman who is pregnant or nursing
3. Patients who have received any stent implantation in the target vessel within one year
4. Patients required long-term oral anticoagulation
5. Known non-adherence to antiplatelet therapy or not suitable for long-term antiplatelet therapy due to high bleeding risk
6. Patients who are allergic to heparin, poly L-lactic acid (PLLA), sirolimus, antiplatelet drugs, or contrast
7. Currently participating in another trial and not yet at its primary endpoint
8. Patients whose life expectancy is less than 3 years
9. Cardiogenic shock

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 36 months
  DoCE is a composite clinical endpoint of cardiovascular death, target vessel myocardial infarction (TV-MI), and clinically and physiologically indicated target lesion revascularization (CPI-TLR).

SECONDARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 1, 12, and 60 months
  Rates of the DoCE beside the time point of primary endpoint
Patient-oriented composite endpoint (PoCE) | 1, 12, 36, and 60 months
  PoCE is defined as a composite endpoint including all-cause death, stroke, myocardial infarction, and revascularization
Target vessel failure (TVF) | 1, 12, 36, and 60 months
  TVF is defined as a composite endpoint including cardiovascular death, TV-MI and clinically and physiologically target vessel revascularization
All-cause death | 1, 12, 36, and 60 months
  Individual components of PoCE
Cardiovascular death | 1, 12, 36, and 60 months
  Individual components of the DoCE
Stroke | 1, 12, 36, and 60 months
  Individual components of PoCE
Myocardial infarction | 1, 12, 36, and 60 months
  Individual components of PoCE
Target vessel myocardial infarction (TV-MI) | 1, 12, 36, and 60 months
  Individual components of DoCE
Revascularization | 1, 12, 36, and 60 months
  Individual components of PoCE
Clinically and physiologically indicated target vessel revascularization | 1, 12, 36, and 60 months
  Individual components of TVF
Clinically and physiologically indicated target lesion revascularization (CPI-TLR) | 1, 12, 36, and 60 months
  Individual components of the DoCE
Definite/Probable scaffold/stent thrombosis | 1, 12, 36, and 60 months
  According to ARC-2 definitions
BARC defined type 3 or 5 bleeding events | 1, 12, 36, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D., Study Chair — Xijing Hospital; Patrick Serruys, M.D., Ph.D., Study Chair — National University of Ireland, Galway; Yoshinobu Onuma, M.D., Ph.D., Study Chair — National University of Ireland, Galway; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No